CLINICAL TRIAL: NCT02760784
Title: Medium Term Outcome of Nonoperative Dynamic Treatment of Acute Achilles Tendon Rupture: the Influence of Early Weight-bearing on Clinical Outcome: a Blinded, Randomized Controlled Trial.
Brief Title: Medium Term Outcome of Nonoperative Treatment After Achilles Tendon Rupture.
Status: Completed | Type: Observational
Sponsor: Copenhagen University Hospital, Hvidovre (Other)
Responsible Party: Principal Investigator, Rasmus Kastoft, Research Assistant, Copenhagen University Hospital, Hvidovre
Other Study IDs: 16015461-1
Record Dates: First submitted 2016-04-25; First posted 2016-05-04 (Estimated); Last update posted 2017-08-10 (Actual); Status verified 2017-08

CONDITIONS: Achilles Tendon Rupture
Keywords: Achilles Tendon Rupture; Conservative treatment; early weight bearing; Dynamic; ATRS; ATRA; Heel Raise Work

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Early Weight Bearing: Ankle immobilized with orthosis (DJO Nextep Contour 2 Walker) with 3 1.5 cm wedges in the heel, fixing the angle between 20-30 degrees. The orthosis was used for 8 weeks, gradually removing the wedges. Full weight bearing was allowed from day 1. The orthosis was worn 24 hours / day the first 2 weeks.
  From week 2 controlled motion exercises and removal of the orthosis 5 times a day.
  Interventions: Behavioral: Early weight bearing
- Control: Ankle immobilized with orthosis (DJO Nextep Contour 2 Walker) with 3 1.5 cm wedges in the heel, fixing the angle between 20-30 degrees. The orthosis was used for 8 weeks, gradually removing the wedges. Weight bearing was allowed from week 6. The orthosis was worn 24 hours / day the first 2 weeks.
  From week 2 controlled motion exercises and removal of the orthosis 5 times a day.

INTERVENTIONS:
Behavioral: Early weight bearing — The intervention implies that the selected patients, will be allowed to bear weight on the injured leg form day 1 while wearing the orthosis, in contrast to the control group, who must wait 6 weaks.
  Groups: Early Weight Bearing

SUMMARY:
A total of 56 patients completed a previous study regarding non-operative treatment for acute achilles tendon rupture. This study consists of an additional follow up after 4-5 years depending on original date of injury.

DETAILED DESCRIPTION:
30 patients suffering from acute Achilles tendon rupture was originally randomized to each arm, and followed up after 6 and 12 months. Of these a total of 56 patients was included in the final analysis, and invited to participate in this additional follow-up, 4-5 years after their original injury. Originally patients was monitored using: ATRS questionnaires, ATRA: Achilles Tendon Resting Angle, Heel Raise Work: number of lifts, lift height and total work, and tests of strength and stiffness in the ankle using a kinetic dynamometer.

ELIGIBILITY:
Inclusion Criteria:

* Suffered acute Achilles tendon rupture from April 2011 to March 2012, and then referred to Copenhagen University Hospital Hvidovre.
* Participated and completed the original study.
* The patient must be able to speak and understand Danish, as well as be capable to give informed consent to participating.

Exclusion Criteria:

* Terminal disease or serious illnesses with an ASA score of 3 or above.
* Any injury significantly influencing gate and function of the lower extremities other than re-rupture of the Achilles tendon.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Patients who participated and completed the original study:
  Barfod, K.W., et al., Nonoperative dynamic treatment of acute achilles tendon rupture: the influence of early weight-bearing on clinical outcome: a blinded, randomized controlled trial. J Bone Joint Surg Am, 2014. 96(18): p. 1497-503.
Sampling Method: Non-Probability Sample
Enrollment: 37 (Actual)
Dates: Start 2016-01; Primary Completion 2016-06 (Actual); Study Completion 2017-08 (Actual)

PRIMARY OUTCOMES:
ATRS: Achilles Tendon Rupture Score | approximate 5 years
  From initial test 6 and 12 months after injury, and now 4-5 years after.

SECONDARY OUTCOMES:
Heel Raise Work | Test is performed once, 4-5 years after the initial injury
  The total work (joules), max height of lift (mm) and number of lifts is recorded. THe patient is placed standing on one leg on a platform tilted 10 degrees (heel below toes), and is asked to lift the heel (and thereby bodyweight) as high as possible, once every 2 seconds. When the patient can no longer maintain height or pace, the test is finished.
return to sport and return to work | 4-5 years after the initial injury
  When did the patients return to work full or part time, and when did they take up sports again.

CONTACTS AND LOCATIONS:
Overall Officials: Jeannette Penny, MD, PhD, Study Director — Copenhagen University Hospital, Hvidovre; Rasmus Kastoft, Stud. Med., Principal Investigator — Copenhagen University Hospital, Hvidovre
Locations (1):
- Hvidovre Hospital, Hvidovre, Outside US/Canada/Australia, Denmark

IPD SHARING:
Plan to Share IPD: No
No plan to share data

REFERENCES:
- [Background] Barfod KW, Bencke J, Lauridsen HB, Ban I, Ebskov L, Troelsen A. Nonoperative dynamic treatment of acute achilles tendon rupture: the influence of early weight-bearing on clinical outcome: a blinded, randomized controlled trial. J Bone Joint Surg Am. 2014 Sep 17;96(18):1497-503. doi: 10.2106/JBJS.M.01273. PMID 25232073
- [Derived] Kastoft R, Barfod K, Bencke J, Speedtsberg MB, Hansen SB, Penny JO. 1.7 cm elongated Achilles tendon did not alter walking gait kinematics 4.5 years after non-surgical treatment. Knee Surg Sports Traumatol Arthrosc. 2022 Oct;30(10):3579-3587. doi: 10.1007/s00167-022-06874-y. Epub 2022 Mar 2. PMID 35234975
- [Derived] Speedtsberg MB, Kastoft R, Barfod KW, Penny JO, Bencke J. Gait Function and Postural Control 4.5 Years After Nonoperative Dynamic Treatment of Acute Achilles Tendon Ruptures. Orthop J Sports Med. 2019 Jun 27;7(6):2325967119854324. doi: 10.1177/2325967119854324. eCollection 2019 Jun. PMID 31276005
- [Derived] Kastoft R, Bencke J, Speedtsberg MB, Penny JO, Barfod K. Early weight-bearing in nonoperative treatment of acute Achilles tendon rupture did not influence mid-term outcome: a blinded, randomised controlled trial. Knee Surg Sports Traumatol Arthrosc. 2019 Sep;27(9):2781-2788. doi: 10.1007/s00167-018-5058-4. Epub 2018 Jul 20. PMID 30030579